CLINICAL TRIAL: NCT05853029
Title: Combined Shockwave Therapy Versus Focused Shockwave Therapy in Patients With Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mennallah Ahmed Mohamed Anwar Elgendy (Other)
Responsible Party: Sponsor-Investigator, Mennallah Ahmed Mohamed Anwar Elgendy, Principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Shockwave on tennis elbow
Record Dates: First submitted 2023-03-26; First posted 2023-05-10 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Epicondylitis
Keywords: Shockwave therapy; Lateral epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Masking Description: Randomization using envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group (1): Twenty patients will receive 2000 pulses of Focused shock wave therapy with (4 Hz; 0.2 millijoule (mJ)/mm2) in addition to conventional therapy including eccentric exercises, stretching, hot packs and deep transverse friction(Johnson et al., 2007). Each patient will have 3 treatment sessions held at weekly basis(Król et al., 2015).
  Interventions: Combination Product: Combined shockwave therapy & conventional therapy , focused shockwave therapy& conventional therapy , conventional therapy
- Group B (Experimental): Group (2): Twenty patients will receive both 2000 pulses of (Focused shockwave therapy with (4 Hz; 0.2 mJ/mm2) and 2000 pulses of Radial shockwave therapy with (8 Hz, 2.5 bars) )= combined shockwave therapy in addition to conventional therapy including eccentric exercises, stretching, hot packs and deep transverse friction(Johnson et al., 2007). Each patient will have 3 treatment sessions held at weekly basis(Król et al., 2015).
  Interventions: Combination Product: Combined shockwave therapy & conventional therapy , focused shockwave therapy& conventional therapy , conventional therapy
- Group C (Experimental): Group (3): Control group of twenty patients that will only receive conventional therapy including eccentric exercises, stretching, hot packs and deep transverse friction(Johnson et al., 2007).
  Interventions: Combination Product: Combined shockwave therapy & conventional therapy , focused shockwave therapy& conventional therapy , conventional therapy

INTERVENTIONS:
Combination Product: Combined shockwave therapy & conventional therapy , focused shockwave therapy& conventional therapy , conventional therapy — The device used for management is from Storz-Medical company; Duolith-SD1 with focused and radial module.
  - Conventional therapy in the form of eccentric exercises, stretching, hot packs and deep transverse friction(Johnson et al., 2007).
  Other Names: Conventional therapy for tennis elbow

SUMMARY:
1. To determine the best effective modality between combined (focused and radial) and focused shockwave therapy for treatment of lateral epicondylitis regarding pain.
2. To determine the best effective modality between combined (focused and radial) and focused shockwave therapy for treatment of lateral epicondylitis regarding hand function.
3. 1. To determine the best effective modality between combined (focused and radial) and focused shockwave therapy for treatment of lateral epicondylitis regarding grip strength.

DETAILED DESCRIPTION:
Lateral epicondylitis, also known as "tennis elbow", is a common disease present in clinical practice. It affects 1% to 3% in the general population which can reach up to 29% in certain occupations with repetitive wrist movements. It can cause a significant functional decline with a great psychological and economic impact.

Major symptoms include decreased grip and upper-extremity strength along with pain and inflammation originating from the lateral elbow. The pathogenesis of lateral epicondylitis is still controversial, but it is known that not only the tendon of the extensor carpi radialis brevis (ECRB) muscle but also the annular ligament, lateral capsule, radial nerve and some bands of the extensor digitorum communis muscle are involved.

It was originally thought that the cause of lateral epicondylitis was an inflammatory process, which would then result in the symptoms. However, histological studies have demonstrated that, through repetitive injuries at this site, there is a degenerative process and a failure of repair in the ECRB tendon. This is more pronounced than inflammation in other structures.

A variety of therapeutic techniques have been proposed for the appropriate management of patients with lateral elbow tendinopathy including exercise, orthotics, manual therapy, passive modalities, acupuncture or a combination of them.

However, the effectiveness of each treatment option remains debatable. Extracorporeal shockwave therapy (ESWT) is a popular method in the management of common tendinopathies and has been proposed as an effective supplement to other non-invasive therapies. There are two types of extracorporeal shockwave therapy: focused shockwave therapy (FSWT) and radial shockwave therapy (RSWT). Waves that are generated for focused and radial ESWT have very different physical characteristics.

FSWT has focused on a pressure area concentrated on a definite place, and can be adjusted at definite depths in the selected tissues, where the higher pressure is touched. Focused type of shockwave is directed by the reflection at definitive areas into the body of patients, and the waves are generated from a wide arc, hence the amount of energy discrete is minimal at the point of real wave generation. The radial shock wave therapy has been attributed to the scattering pressure zone of RSWT apparatus, which arrives at the source as the highest pressure, and didn't require a certain distance in human body and the omitted waves radiate within the tissues, and influence a large area, but they do not deeply reach the thick tissues as that in focused wave therapy, therefore RSWT is effective for treating superficial lesions that assist the deep-tissue stimulation like backs and muscles.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 18 - 55 years old.
* BMI < 35
* Males and Females
* Painful chronic tennis elbow during at least 3 previous months identified by positive Mill"s, Maudsley"s and Cozen"s tests.
* Painful palpation of the lateral epicondyle.
* Painful resisted middle finger and wrist extension (Maudsley's test).

Exclusion Criteria:

* Local infection.
* Malignancy.
* Elbow arthritis or instability.
* Pronator-Teres syndrome.
* Generalized polyarthritis.
* Neurological disorders (Stroke and Parkinson"s disease).
* Radial-nerve entrapment.
* Physical therapy and/or a corticosteroid injection administered within the previous six weeks.
* Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Visual analog Scale (VAS) for pain to will be carried out for each patient individually before, immediately after treatment and 2 months after end of treatment. | 3 months
  amount of pain the VAS scale will be employed, where 0 indicates "no pain" and 10 indicates "most severe pain
rated-tennis-elbow-questionnaire for hand function assessment | 3 months
  score from that questionnaire Pain Subscale - Add up 5 items. Best score = 0; Worst score = 50 Specific Activities - Add up 6 items Best Score = 0; Worst Score = 60 Usual Activities - Add up 4 items items Best Score = 0; Worst Score = 40 Function Subscale - (Specific Activities + Usual Activities) /2 Best score = 0; Worst score = 50 Total Score = Pain Subscale + Function Subscale Best Score = 0; Worst Score = 100 (pain and disability contribute equally to score)
Grip strength will be measured using the CAMRY digital hand dynamometer, model EH101 | 3 months
  Device used to test the hand grib strength

SECONDARY OUTCOMES:
For patient selection Mill's Test | Before the study for patient selection
  Patient's lateral epicondyle palpated with one hand, while pronating the patient's forearm, fully flexing the wrist, the elbow extended. Decided it a positive test when we found pain in the area of insertion at lateral epicondyle.
Maudsley's test | Before the study for patient selection
  The examiner resists extension of the 3rd digit of the hand, stressing the extensor digitorum muscle and tendon, while palpating the patient's lateral epicondyle. A positive test is indicated by pain over the lateral epicondyle of the humerus.
Cozen's Test | Before the study for patient selection
  To perform Cozen's test,patient seated, the therapist stabilizes the patient's elbow in 90 degrees of flexion with one hand while palpating over the lateral epicondyle. The other hand positions the patient's hand into radial deviation and forearm pronation while the patient is asked to resisted wrist extension in this position against manual resistance of the therapist. The test is considered positive if it produces pain or reproduction of other symptoms in the area of the lateral epicondyle.

CONTACTS AND LOCATIONS:
Overall Officials: RANIA REDA, A. Prof Dr., Study Director — cairo uni; NEVEEN Abdelraoof, Prof. Dr., Study Director — cairo uni; Menna allah Elgendy, Bachelor, Principal Investigator — cairo uni; Titus Bertolini, Dr. med., Study Director — Medicum clinics Germany

REFERENCES:
- [Background] Levin D, Nazarian LN, Miller TT, O'Kane PL, Feld RI, Parker L, McShane JM. Lateral epicondylitis of the elbow: US findings. Radiology. 2005 Oct;237(1):230-4. doi: 10.1148/radiol.2371040784. Epub 2005 Aug 18. PMID 16118152
- [Background] Aben A, De Wilde L, Hollevoet N, Henriquez C, Vandeweerdt M, Ponnet K, Van Tongel A. Tennis elbow: associated psychological factors. J Shoulder Elbow Surg. 2018 Mar;27(3):387-392. doi: 10.1016/j.jse.2017.11.033. PMID 29433642
- [Background] Abo Al-Khair MA, El Khouly RM, Khodair SA, Al Sattar Elsergany MA, Hussein MI, Eldin Mowafy ME. Focused, radial and combined shock wave therapy in treatment of calcific shoulder tendinopathy. Phys Sportsmed. 2021 Nov;49(4):480-487. doi: 10.1080/00913847.2020.1856633. Epub 2020 Dec 6. PMID 33283581
- [Background] Baker CL Jr, Baker CL 3rd. Long-term follow-up of arthroscopic treatment of lateral epicondylitis. Am J Sports Med. 2008 Feb;36(2):254-60. doi: 10.1177/0363546507311599. PMID 18202296
- [Background] Bisset LM, Vicenzino B. Physiotherapy management of lateral epicondylalgia. J Physiother. 2015 Oct;61(4):174-81. doi: 10.1016/j.jphys.2015.07.015. Epub 2015 Sep 8. No abstract available. PMID 26361816
- [Background] Chang KV, Chen SY, Chen WS, Tu YK, Chien KL. Comparative effectiveness of focused shock wave therapy of different intensity levels and radial shock wave therapy for treating plantar fasciitis: a systematic review and network meta-analysis. Arch Phys Med Rehabil. 2012 Jul;93(7):1259-68. doi: 10.1016/j.apmr.2012.02.023. Epub 2012 Mar 12. PMID 22421623
- [Background] Cohen M, da Rocha Motta Filho G. LATERAL EPICONDYLITIS OF THE ELBOW. Rev Bras Ortop. 2015 Dec 8;47(4):414-20. doi: 10.1016/S2255-4971(15)30121-X. eCollection 2012 Jul-Aug. PMID 27047843
- [Background] Hastie G, Soufi M, Wilson J, Roy B. Platelet rich plasma injections for lateral epicondylitis of the elbow reduce the need for surgical intervention. J Orthop. 2018 Jan 31;15(1):239-241. doi: 10.1016/j.jor.2018.01.046. eCollection 2018 Mar. PMID 29657476
- [Background] Gerdesmeyer L, Frey C, Vester J, Maier M, Weil L Jr, Weil L Sr, Russlies M, Stienstra J, Scurran B, Fedder K, Diehl P, Lohrer H, Henne M, Gollwitzer H. Radial extracorporeal shock wave therapy is safe and effective in the treatment of chronic recalcitrant plantar fasciitis: results of a confirmatory randomized placebo-controlled multicenter study. Am J Sports Med. 2008 Nov;36(11):2100-9. doi: 10.1177/0363546508324176. Epub 2008 Oct 1. PMID 18832341
- [Background] Ilieva EM, Minchev RM, Petrova NS. Radial shock wave therapy in patients with lateral epicondylitis. Folia Med (Plovdiv). 2012 Jul-Sep;54(3):35-41. doi: 10.2478/v10153-011-0095-5. PMID 23270205
- [Background] Karanasios S, Tsamasiotis GK, Michopoulos K, Sakellari V, Gioftsos G. Clinical effectiveness of shockwave therapy in lateral elbow tendinopathy: systematic review and meta-analysis. Clin Rehabil. 2021 Oct;35(10):1383-1398. doi: 10.1177/02692155211006860. Epub 2021 Apr 4. PMID 33813913
- [Background] Korakakis V, Whiteley R, Tzavara A, Malliaropoulos N. The effectiveness of extracorporeal shockwave therapy in common lower limb conditions: a systematic review including quantification of patient-rated pain reduction. Br J Sports Med. 2018 Mar;52(6):387-407. doi: 10.1136/bjsports-2016-097347. Epub 2017 Sep 27. PMID 28954794
- [Background] Krol P, Franek A, Durmala J, Blaszczak E, Ficek K, Krol B, Detko E, Wnuk B, Bialek L, Taradaj J. Focused and Radial Shock Wave Therapy in the Treatment of Tennis Elbow: A Pilot Randomised Controlled Study. J Hum Kinet. 2015 Oct 14;47:127-35. doi: 10.1515/hukin-2015-0068. eCollection 2015 Sep 29. PMID 26557197
- [Background] Lian J, Mohamadi A, Chan JJ, Hanna P, Hemmati D, Lechtig A, Nazarian A. Comparative Efficacy and Safety of Nonsurgical Treatment Options for Enthesopathy of the Extensor Carpi Radialis Brevis: A Systematic Review and Meta-analysis of Randomized Placebo-Controlled Trials. Am J Sports Med. 2019 Oct;47(12):3019-3029. doi: 10.1177/0363546518801914. Epub 2018 Oct 31. PMID 30380334
- [Background] Savoie FH 3rd, VanSice W, O'Brien MJ. Arthroscopic tennis elbow release. J Shoulder Elbow Surg. 2010 Mar;19(2 Suppl):31-6. doi: 10.1016/j.jse.2009.12.016. PMID 20188266
- [Background] Maloney MD, Mohr KJ, el Attrache NS. Elbow injuries in the throwing athlete. Difficult diagnoses and surgical complications. Clin Sports Med. 1999 Oct;18(4):795-809. doi: 10.1016/s0278-5919(05)70185-x. PMID 10553236
- [Background] Nowotny J, El-Zayat B, Goronzy J, Biewener A, Bausenhart F, Greiner S, Kasten P. Prospective randomized controlled trial in the treatment of lateral epicondylitis with a new dynamic wrist orthosis. Eur J Med Res. 2018 Sep 15;23(1):43. doi: 10.1186/s40001-018-0342-9. PMID 30219102
- [Background] Sanders TL Jr, Maradit Kremers H, Bryan AJ, Ransom JE, Smith J, Morrey BF. The epidemiology and health care burden of tennis elbow: a population-based study. Am J Sports Med. 2015 May;43(5):1066-71. doi: 10.1177/0363546514568087. Epub 2015 Feb 5. PMID 25656546
- [Background] Shiri R, Viikari-Juntura E. Lateral and medial epicondylitis: role of occupational factors. Best Pract Res Clin Rheumatol. 2011 Feb;25(1):43-57. doi: 10.1016/j.berh.2011.01.013. PMID 21663849
- [Background] De Smedt T, de Jong A, Van Leemput W, Lieven D, Van Glabbeek F. Lateral epicondylitis in tennis: update on aetiology, biomechanics and treatment. Br J Sports Med. 2007 Nov;41(11):816-9. doi: 10.1136/bjsm.2007.036723. Epub 2007 Jul 6. PMID 17616547
- [Background] Smith AR Jr. Manual therapy: the historical, current, and future role in the treatment of pain. ScientificWorldJournal. 2007 Feb 2;7:109-20. doi: 10.1100/tsw.2007.14. PMID 17334604
- [Background] Spacca G, Necozione S, Cacchio A. Radial shock wave therapy for lateral epicondylitis: a prospective randomised controlled single-blind study. Eura Medicophys. 2005 Mar;41(1):17-25. PMID 16175767
- [Background] Speed C. A systematic review of shockwave therapies in soft tissue conditions: focusing on the evidence. Br J Sports Med. 2014 Nov;48(21):1538-42. doi: 10.1136/bjsports-2012-091961. Epub 2013 Aug 5. PMID 23918444
- [Background] Stania M, Krol B, Franek A, Blaszczak E, Dolibog P, Polak A, Dolibog P, Durmala J, Krol P. A comparative study of the efficacy of radial and focused shock wave therapy for tennis elbow depending on symptom duration. Arch Med Sci. 2020 Apr 6;17(6):1686-1695. doi: 10.5114/aoms.2019.81361. eCollection 2021. PMID 34900050
- [Background] van der Worp H, Zwerver J, Hamstra M, van den Akker-Scheek I, Diercks RL. No difference in effectiveness between focused and radial shockwave therapy for treating patellar tendinopathy: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2014 Sep;22(9):2026-32. doi: 10.1007/s00167-013-2522-z. Epub 2013 May 12. PMID 23666379
- [Background] Yoon SY, Kim YW, Shin IS, Kang S, Moon HI, Lee SC. The Beneficial Effects of Eccentric Exercise in the Management of Lateral Elbow Tendinopathy: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Sep 1;10(17):3968. doi: 10.3390/jcm10173968. PMID 34501416